CLINICAL TRIAL: NCT01623739
Title: Esthetic, Clinical and Radiographic Outcomes of Immediately Placed Implants (Type 1) and Early Placed Implants (Type 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITI 689_2010
Record Dates: First submitted 2012-04-26; First posted 2012-06-20 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2017-10

CONDITIONS: Jaw, Edentulous, Partially; Acquired Absence of Single Tooth
Keywords: Dental implants; Esthetic score; Immediate implants; Early placement
MeSH Terms: conditions — Jaw, Edentulous, Partially | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Type 1 implant placement (Active Comparator): Placement of a dental implant: Implant is placed immediately following tooth extraction in one surgical procedure
  Interventions: Procedure: Placement of a dental implant
- Type 2 implant placement (Active Comparator): Placement of a dental implant: Once the tooth is extracted. The site is left to heal for 4 to 8 weeks before a dental implant is placed during a second surgical procedure.
  Interventions: Procedure: Placement of a dental implant

INTERVENTIONS:
Procedure: Placement of a dental implant — Type 1 implant placement Type 2 implant placement
  Other Names: Straumann; SLActive; Dental Implants

SUMMARY:
The investigators are asking subjects to take part in a research study of soft tissue (gums) and bone (jawbone) healing around dental implants following tooth extraction. The investigators want to compare how the gums and the bone changes shape with healing in two different scenarios:

1. When the implant is placed at the same time the tooth is extracted.
2. When the tooth is extracted and then left to heal for a period of 4 to 8 weeks before the implant is placed.

Previous studies have shown that both methods work and can give good results. In fact the two methods are used routinely as part of standard care but it is not known if the two procedures are equally good since they have never been compared in one same research study.

DETAILED DESCRIPTION:
This controlled, randomized clinical trial (RCT) is designed to compare soft and hard tissue dimensional changes for two commonly used approaches for replacing a recently extracted tooth by means of a dental implant, i.e. immediate implant placement (Type 1) or early implant placement (Type 2). Additionally, this study will evaluate the association between the osseous anatomy and implant position with soft and hard tissue changes.

Extraction sites will include maxillary and mandibular anterior and premolar teeth having intact adjacent teeth. Implants placed for this study will be SLA surface, bone level design, Straumann BL RC (Bone Level Regular Cross-fit ) 4.1mm or BL NC (Bone Level Narrow Cross-fit ) 3.3mm diameter implants at 8, 10, 12 or 14mm in length.

Immediate implant placement (Type 1) resulting in a horizontal defect dimension (HDD) will receive bone grafting, using freeze dried bone allograft (FDBA)(Straumann Allograft GC®) and will be covered by a resorbable membrane (BioGide®).

For the implants randomized to type 2 implant placement, the extraction socket will be filled with a collagen plug and allowed to heal for 4 to 8 weeks before the implant will be placed. Simultaneous guided bone regeneration (GBR) will be performed using FDBA (Straumann Allograft GC®)and a resorbable collagen membrane (BioGide®). The type 2 implant placement procedure will follow the guidelines as described by Buser et al. (2008).

All implant placement will follow standard protocols utilizing tapping and placement according to the manufacturer's guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is 18 years or older.
2. Ability to understand and provide informed consent before starting the study.
3. Ability and willingness to comply with all study requirements.
4. The patient, if of child-bearing potential, has a negative urine pregnancy test.
5. Adequate oral hygiene to allow for implant therapy consistent with standards of care.
6. Adequate bone volume to accommodate the planned endosseous dental implant placement following immediate placement protocols utilizing Straumann Bone Level implants RC 4.1mm or Bone Level Implant NC 3.3 mm at 8, 10, 12 or 14 mm in length.
7. One or more teeth in either the maxilla or mandible anterior or premolar areas requiring extraction leading to a single-tooth gap requiring implant placement as determined by the patient's dental provider.
8. Following extraction, surgical site anatomy presents conditions allowing immediate implant placement.
9. Primary stability of implant consistent with standards of care is achieved at the time of placement.

Exclusion Criteria:

1. Patient reports current smoking habit with moderate or heavy smoking (more than 10 cigarettes per day) or tobacco chewing use.
2. History of alcoholism or drug abuse within the past 5 years.
3. Severe bruxism or clenching habits.
4. Patient has significant untreated periodontal disease (grade III or IV), caries, or clinical or radiographic signs of infection within two adjacent tooth positions of implant area.
5. History of HIV infection, Hepatitis B or C.
6. Patients with a history of systemic disease that precludes standard dental implant therapy or alters daily activities to a level consistent with ASA III classification (including cardiovascular, hepatic, renal, gastrointestinal, metabolic, neurologic, pulmonary, endocrine, autoimmune, or psychiatric disorders).
7. Presence of local inflammation or mucosal diseases such as lichen planus
8. Patient history consistent with high risk for subacute bacterial endocarditis
9. Current hematological disorder or coumadin (or similar) therapy
10. Patient has a disease that affects bone metabolism, such as but not limited to osteoporosis, hyperthyroidism, hyperparathyroidism, congenital connective tissue disorders (e.g., osteogenesis imperfecta), or Paget's disease.
11. Patient is taking medications or having treatments known to have an effect on bone turnover, including: thiazide diuretics, calcitonin, systemic steroids, bisphosphonates, vitamin D (>800 IU/day), estrogen or progesterone therapy.
12. Current steroid treatment: defined as any person who within the last two years has received for two weeks a dose equivalent to 20 mg hydrocortisone
13. Patient currently undergoing chemotherapy
14. Patient history of radiation treatment to the head or neck
15. Physical or mental handicaps that would interfere with patient's ability to exercise good oral hygiene on a regular basis
16. Use of any investigational drug or device within the 30 day period immediately prior to implant surgery
17. Patient is pregnant
18. Extraction sites having anatomic conditions that preclude immediate implant placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Huynh-Ba, DDS, MS, Principal Investigator — UTHSCSA Department of Periodontics
Locations (1):
- Graduate Periodontics, Dental School, UTHSCSA, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Type 1 Implant Placement: Implant is placed immediately following tooth extraction in one surgical procedure
  Placement of a dental implant: Type 1 implant placement Type 2 implant placement
- Type 2 Implant Placement: Once the tooth is extracted. The site is left to heal for 4 to 8 weeks before a dental implant is placed during a second surgical procedure.
  Placement of a dental implant: Type 1 implant placement Type 2 implant placement
Period: Overall Study
Arm/Group | Type 1 Implant Placement | Type 2 Implant Placement
Started | 19 | 19
Completed | 17 | 15
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Type 1 Implant Placement | Type 2 Implant Placement | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (15.6) | 50.9 (14.6) | 51.8 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 9 | 9 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Mid Facial Mucosal Level at Implant Site
Description: Baseline will be at the time of crown delivery. Thereafter, the mid facial mucosal level at implant site will be recorded at 3, 6, 12, 24, 36, 48, 60 months after crown delivery.
Time Frame: 3 months after crown delivery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Type 1 Implant Placement | Type 2 Implant Placement
Number analyzed (Participants) | 17 | 15
mm | 0.54 (0.18) | 0.47 (0.31)

2. Secondary Outcome: PES/WES (Pink Esthetic Score, White Esthetic Score).
Description: The PES and WES scales are 10 point scales, made up of 5 categories, each with a 2 point value. Each category is scored out of 2, and the scores totaled to give an optimal score out of 10. Any score of 6 or higher out of 10 would be considered a good clinical outcome. the PES categories focus on the gum area, and the WES categories focus on the tooth. The scores for PES and WES are totaled, to give a score out of 20, with 20 being the highest possible score (best outcome). The values are totaled and a mean score of all the readings is reported.
Time Frame: 3, 6, 12, 24, 36, 48, 60 months after crown delivery
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Type 1 Implant Placement | Type 2 Implant Placement
Number analyzed (Participants) | 17 | 15
units on a scale | 13.67 (0.61) | 12.51 (0.65)

3. Secondary Outcome: Probing Depth
Description: The measurement of the pocket around the implanted tooth, measured with a graduated probe. A healthy pocket depth is around 3mm with no bleeding during the measurement process. The values are totaled and a mean score of all the readings is reported.
Time Frame: 3, 6, 12, 24, 36, 48, 60 months after crown delivery
Measure: Mean (Standard Error); unit: mm
Arm/Group | Type 1 Implant Placement | Type 2 Implant Placement
Number analyzed (Participants) | 17 | 15
mm | 3.06 (0.18) | 2.93 (0.18)

4. Secondary Outcome: Modified Plaque Index
Description: Measurement of amount of plaque build-up on teeth, using a scale of 0 (no plaque detection), to 3 (an abundance of soft matter). The scores are totaled and a mean score reported.
Time Frame: 3, 6, 12, 24, 36, 48, 60 months after crown delivery
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Type 1 Implant Placement | Type 2 Implant Placement
Number analyzed (Participants) | 17 | 15
units on a scale | 0.18 (0.10) | 0.27 (0.15)

5. Secondary Outcome: Modified Bleeding Index
Description: Bleeding from the gums is measured on probing the gum and measured on scale of 0 to 5, with 0 being the best outcome, with no bleeding, and 5 being the worst outcome, with spontaneous bleeding. The scores are totaled and a mean score reported.
Time Frame: 3, 6, 12, 24, 36, 48, 60 months after crown delivery
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Type 1 Implant Placement | Type 2 Implant Placement
Number analyzed (Participants) | 17 | 15
units on a scale | 0.12 (0.08) | 0.07 (0.07)

6. Secondary Outcome: Radiographic Bone Level
Description: Secondary outcome measures will be recorded at 3, 6, 12, 24, 36, 48, 60 months after crown delivery.
Time Frame: Up to 5 years after baseline
Population: No data were collected or analyzed for this outcome measure
Groups:
- Radiographic Bone Level: Radiography is used to measure amount of bone
Arm/Group | Radiographic Bone Level
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 3 months after crown delivery
Arm/Group | Type 1 Implant Placement | Type 2 Implant Placement
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/17 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type 1 Implant Placement (N=17) | Type 2 Implant Placement (N=15)
Swelling and bruising (Surgical and medical procedures) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No